CLINICAL TRIAL: NCT00599040
Title: The DINE Study-Diet Intervention to Negate Diabetes Study (Improving Weight Loss Outcomes for African Americans)
Acronym: DINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jamy Ard, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: F040719005; 1K23DK068223-01 (NIH)
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes; Hypertension; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Weight loss (Active Comparator): Weight loss diet focused on the DASH diet
  Interventions: Behavioral: The DASH diet with weight loss
- DASH diet (Active Comparator): The DASH diet without weight loss
  Interventions: Behavioral: The DASH diet without weight loss
- Diary (Active Comparator): Dairy Intervention
  Interventions: Behavioral: Dairy diet

INTERVENTIONS:
Behavioral: The DASH diet with weight loss — A reduced calorie diet is provided to participants based on the DASH diet.
  Arms: Weight loss
Behavioral: The DASH diet without weight loss — participants are given a weight maintainenance diet based on the DASH diet
  Arms: DASH diet
Behavioral: Dairy diet — participants are given a high dairy, reduced calorie diet
  Arms: Diary

SUMMARY:
The purpose of this study is to determine if what you eat affets your insulin sensitivity when you lose a small amount of weight

ELIGIBILITY:
Inclusion Criteria:

* African American adults (age ≥ 19)
* Obese (BMI > or equal to 30 kg/m2)
* Otherwise generally healthy

Exclusion Criteria:

* Diagnoses of diabetes
* Malignancy or other states where weight loss is contraindicated (pregnancy
* Individuals with high blood pressure on medications.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jamy D Ard, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Nutrition Sciences Department, Birmingham, Alabama, United States